CLINICAL TRIAL: NCT05023486
Title: NP-G2-044 as Monotherapy and Combination Therapy in Patients With Advanced or Metastatic Solid Tumor Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novita Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP-G2-044-P2-01
Record Dates: First submitted 2021-07-30; First posted 2021-08-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-08

CONDITIONS: Advanced or Metastatic Solid Tumor Malignancies
Keywords: Advanced or Metastatic Solid Tumor Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NP-G2-044 Monotherapy - Capsule/Tablet (Experimental): NP-G2-044 capsule/tablet PO QD for each 28-day cycle
  Interventions: Drug: NP-G2-044 Monotherapy
- NP-G2-044 Combination Therapy With Anti-PD-1 Therapy (Experimental): NP-G2-044 capsules PO QD for each 28-day cycle, Anti-PD-1 Therapy per standard of care, at a dose and frequency in accordance with the package insert
  Interventions: Drug: Anti-PD-1 Therapy; Drug: NP-G2-044 Combination therapy

INTERVENTIONS:
Drug: NP-G2-044 Monotherapy — 1600 mg QD, 2000mg QD, and 2100 mg QD
  Arms: NP-G2-044 Monotherapy - Capsule/Tablet
Drug: Anti-PD-1 Therapy — previously initiated per standard of care, at a dose and frequency in accordance with the package insert
  Arms: NP-G2-044 Combination Therapy With Anti-PD-1 Therapy
Drug: NP-G2-044 Combination therapy — 1600 mg QD or 2100 mg QD
  Arms: NP-G2-044 Combination Therapy With Anti-PD-1 Therapy

SUMMARY:
Multicenter, open-label study in patients with advanced or metastatic solid tumor malignancies to evaluate the safety, tolerability, and preliminary anti-tumor efficacy, PK, and pharmacodynamics of continuously dosed NP-G2-044 monotherapy and NP-G2-044 in combination with anti-PD-1 therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 years of age;
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
3. Life expectancy of > 6 months;
4. Abilty to swallow capsules and tablets;
5. Adequate organ and bone marrow function, defined by the following:

   ANC >1500 cells/μL; Hemoglobin >9.0 g/dL; Platelet count >100,000 cells/μL; Total bilirubin ≤1.5 mg/dL; Albumin ≥3.0 g/dL; Alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, and gamma-glutamyl transferase ≤2.5 × upper limit of normal (ULN); Creatinine clearance ≥50 mL/min; and Prothrombin time and partial thromboplastin time ≤1.5 × ULN.
6. Female patients of childbearing potential must have a negative serum or urine pregnancy test at Screening and within 24 hours (if urine test) or 72 hours (if serum test) before the first dose of NP-G2-044. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required and must be negative for the patient to be eligible; Note: A woman is considered to be childbearing potential unless she is postmenopausal (≥1 year without menses and confirmed with a follicle-stimulating hormone [FSH] test) or surgically sterilized via bilateral oophorectomy, hysterectomy, bilateral tubal ligation, or successful Essure® placement with a documented confirmation test at least 3 months after the procedure.
7. Male patients must be surgically sterile or willing to use a highly effective double-barrier contraception method (e.g., male condom with diaphragm or male condom with cervical cap) upon study entry, while on NP-G2-044, and for a period of at least 4 months following the last dose of NP-G2-044; and
8. Able to understand and voluntarily sign a written informed consent form (ICF) and willing and able to comply with protocol requirements.

Inclusion Criteria for NP-G2-044 Monotherapy:

Patients must meet all the following criteria to receive NP-G2-044 monotherapy in the study:

1. Have a histopathologically confirmed advanced or metastatic solid tumor malignancy for which standard therapies are no longer effective, not tolerated or ineligible for the patient to receive;
2. Have measurable disease per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1);
3. For monotherapy expansion cohort A (after the Mono-RP2D has been identified), patients must have:

   1. Gynecologic malignancies including ovarian, endometrial/uterine, fallopian tube, cervical, vulvar, and vaginal cancers; or
   2. Epidermal growth factor receptor (EGFR)-high (2+ or 3+ staining per DAKO criteria or genomic sequencing data showing 3 or more copies of the EGFR gene) triple-negative breast cancer (TNBC).
4. For Monotherapy Expansion Cohort B, patient must have advanced or metastatic solid tumors malignancy

Inclusion Criteria for NP-G2-044 Combination Therapy Patients must meet the following criteria to receive NP-G2-044 in combination with anti-PD-1 therapy in the study:

1. Have measurable disease per RECIST 1.1;

   For Combination Therapy Expansion Cohort A:
2. Patients must meet 1 of the following criteria to enroll in Combination Therapy Expansion Cohort A:

   1. Have initiated anti-PD-(L)1 therapy in accordance with the package insert and have been receiving the anti-PD-(L)1 therapy for ≥3 months (with therapy currently ongoing) and have stable disease (defined either by post-treatment onset radiographic scan or ≥3 months without radiographic or clinical evidence of progression), or had an initial period of stable disease and now have an initial scan demonstrating progressive disease per RECIST 1.1. or
   2. Have discontinued prior anti-PD-(L)1 therapy and are now eligible for de novo NP-G2-044 plus standard of care anti-PD-1 therapy.

   For Combination Therapy Expansion Cohorts B through E:
3. Patients must meet 1 of the following criteria to enroll in Combination Therapy Expansion Cohorts B through E:

   1. Have initiated anti-PD-(L)1 therapy. in accordance with the package insert and have been receiving the anti-PD-(L)1 therapy for >3 months (with therapy currently ongoing) and have stable disease (as defined above), or had an initial period of stable disease or response and now have an initial scan demonstrating progressive disease per RECIST 1.1; or
   2. Have confirmed progressive disease and discontinued prior anti-PD-(L)1 therapy and are now eligible for de novo NP-G2-044 plus standard of care anti-PD-1 therapy.
4. For Combination Therapy Expansion Cohort B, patients must have cutaneous squamous cell carcinoma (CSCC) (human papilloma virus [HPV]-positive or -negative; documentation of HPV status is required);
5. For Combination Therapy Expansion Cohort C, patients must have either:

   1. Esophageal squamous cell carcinoma (ESCC) (HPV-positive or -negative; documentation of HPV status is required); or
   2. Oropharyngeal squamous cell carcinoma (OPSCC) (HPV-positive or -negative; documentation of HPV status is required).
6. For Combination Therapy Expansion Cohort D, patients must have non muscle invasive bladder cancer (NMIBC) meeting Bacillus Calmette-Guérin (BCG)-unresponsive criteria;
7. For Combination Therapy Expansion Cohort E, patients must have microsatellite instability high (MSI-H) cancer;

   For Combination Therapy Expansion Cohorts F and G:
8. For Combination Therapy Expansion Cohort F, patients must be immunotherapy naïve (I O naïve), have pancreatic ductal adenocarcinoma (PDAC), and meet the following criteria:

   1. Have had stable disease or response with at least 4 months of standard of care chemotherapy;
   2. Have no liver metastasis; and
   3. Have albumin within the normal range at Screening and >3.5 g/dL (±10%) 3 days before Cycle 1 Day 1.
9. For Combination Therapy Expansion Cohort G, patients must be I O naïve, have platinum resistant ovarian cancer (PROC), and meet the following criteria:

   1. Had disease recurrence during or within 6 months after last administration of platinum-based chemotherapy; and
   2. Received no more than 2 prior regimens of systemic therapy after development of platinum resistance.

Exclusion Criteria:

1. Received chemotherapy or radiotherapy within 4 weeks or 5 half-lives, whichever is shorter, of the first dose of NP-G2-044; Note: Prior immunotherapy is allowed for patients receiving NP-G2-044 monotherapy. For PDAC patients in Combination Therapy Expansion Cohort F: received systemic therapy within 2 weeks of the first dose of NP-G2-044.
2. Unresolved toxicities from previous anti-cancer therapy, defined as toxicities (other than NCI CTCAE v5.0 Grade ≤2 alopecia or neuropathy) not yet resolved to NCI CTCAE v5.0 Grade ≤1; Note: Patients who experienced a Grade ≥3 anti-PD-1-related AE per NCI CTCAE v5.0 are excluded unless recovered and approved by the Novita Medical Monitor or designee.
3. Receiving any other investigational agent(s) or have received an investigational agent within 4 weeks of the first dose of NP-G2-044; Note: Patients who have progressed on NP-G2-044 treatment prior to this study are not eligible
4. Known untreated brain metastases or treated brain metastases that have not been radiographically and clinically stable (i.e., not requiring steroids) ≥4 weeks prior to study enrollment;
5. QTc by Fridericia method >470 msec or electrocardiogram (ECG) with evidence of clinically meaningful conduction abnormalities or active ischemia as determined by the Investigator;
6. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, hypertension, unstable angina pectoris, cardiac arrhythmia, autoimmune or inflammatory diseases, or psychiatric illness/social situations that would limit compliance with study requirements;
7. Pregnant, lactating, or is planning to attempt to become pregnant or impregnate someone during the study or within 90 days after dosing of NP-G2-044;
8. Received prior allogenic hematopoietic stem cell transplantation or allogenic bone marrow transplantation;
9. Received prior solid organ transplantation;
10. Ongoing immunosuppressive therapy (≥10 mg/day of prednisone or its equivalent);
11. Requires the use of a strong inhibitor or inducer of cytochrome P450 (CYP)3A4, CYP1A2, or CYP2D6 during the study;
12. History of clinically meaningful gastrointestinal bleeding, intestinal obstruction, or gastrointestinal perforation within 6 months of study enrollment;
13. Excluded by the Sponsor due to medical history, physical examination findings, clinical laboratory results, prior medications, or other entrance criteria; or
14. For PDAC patients in Combination Therapy Expansion Cohort F only: have a documented rise in tumor markers within the last 4 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-12-07 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Identification of the NP-G2-044 Monotherapy Recommended Phase 2 Dose (RP2D) | 6 months
Number of incidences of Treatment Emergent Adverse Events with NP-G2-044 monotherapy | Time of first dose of any study drug(s) until 30 days after the last dose of study drug(s)
  Will use NCI CTCAE v5.0
NP-G2-044 anti-tumor preliminary efficacy signals when administered as continuously dosed monotherapy assessed by RECIST 1.1 | 24 months
  (computed tomography [CT] or magnetic resonance imaging [MRI])
Identification of the RP2D for patients receiving NP-G2-044 in combination with anti-PD-1 therapy | 9 months
Number of incidences of Treatment Emergent Adverse Events with NP-G2-044 and anti-PD-1 combination therapy | Time of first dose of any study drug(s) until 30 days after the last dose of study drug(s)
  Will use NCI CTCAE v5.0
NP-G2-044 anti-tumor preliminary efficacy signals when administered in combination with anti-PD-1 therapy assessed by RECIST 1.1 | 24 months
  (computed tomography [CT] or magnetic resonance imaging [MRI])

SECONDARY OUTCOMES:
Identify and characterize preliminary anti-tumor activity of NP-G2-044 in combination with anti-PD-1 therapy | 24 months
  Anti-tumor activity assessed using iRECIST
Pharmacokinetics (PK) of NP-G2-044 monotherapy: AUC | 6 months
  Area under the plasma concentration versus time curve
Pharmacokinetics (PK) of NP-G2-044 monotherapy: Tmax | 6 months
  Time to peak plasma concentration
Pharmacokinetics (PK) of NP-G2-044 monotherapy: Cmax | 6 months
  Peak plasma concentration
Pharmacokinetics (PK) of NP-G2-044 and anti-PD-1 Combination therapy: AUC | 9 months
  Area under the plasma concentration versus time curve
Pharmacokinetics (PK) of NP-G2-044 and anti-PD-1 Combination therapy: Tmax | 9 months
  Time to peak plasma concentration
Pharmacokinetics (PK) of NP-G2-044 and anti-PD-1 Combination therapy: Cmax | 9 months
  Peak plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Zhang, Ph.D., Study Director — Novita Pharmaceuticals, Inc.
Locations (18):
- United States (18):
  - Honor Health Research Institute, Scottsdale, Arizona
  - University of Arizona - Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - City of Hope Irvine Lennar, Irvine, California
  - Hoag Memorial Hospital Presbyterian - Gynecologic Oncology Associates, Newport Beach, California
  - Nuvance Health, Norwalk, Connecticut
  - University of Florida (UF) - Shands Cancer Center, Gainesville, Florida
  - Indiana University (IU) Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Cancer Center, Fairway, Kansas
  - Henry Ford Health System, Detroit, Michigan
  - Atlantic Health System - Morristown Medical Center, Morristown, New Jersey
  - University of Cincinnati (UC) - Cancer Institute, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Commonwealth University - Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No